CLINICAL TRIAL: NCT02929446
Title: Postoperative Mobilization Immediate After Open Abdominal Surgery
Brief Title: Mobilization Immediate After Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Nygren-Bonnier, RPT, PhD, Senior lecturer, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIDAS
Record Dates: First submitted 2016-10-05; First posted 2016-10-11 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Insufficiency; Postoperative Pulmonary Complications
Keywords: mobilisation; physiotherapy
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The interventions were not possible to mask for patients or healthcare professionals at the recovery unit. The research nurses and the physiotherapists, who performed the postoperative spirometry, were blinded to the group randomization. All data were coded, and group assignment was blinded for outcome analyses
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mobilisation (Experimental): Mobilisation out of bed to sit in an armchair or on the bedside, instructed to sit as long as possible
  Interventions: Procedure: Mobilisation
- Control (No Intervention): No mobilisation or breathing exercises until discharge or maximum 6 hours
- Mobilisation and breathing exercises (PEP) (Experimental): Mobilisation out of bed to sit in an armchair or on the bedside, instructed to sit as long as possible and breathing exercises with PEP
  Interventions: Procedure: Mobilisation and breathing exercises

INTERVENTIONS:
Procedure: Mobilisation — Mobilisation out of bed to sit in an armchair or on the bedside, instructed to sit as long as possible
  Arms: Mobilisation
Procedure: Mobilisation and breathing exercises — Mobilisation out of bed to sit in an armchair or on the bedside, instructed to sit as long as possible and breathing exercises with PEP
  Arms: Mobilisation and breathing exercises (PEP)

SUMMARY:
Advances in surgical technique have led to a more complex surgery on patients with more serious comorbidities and the risk of postoperative pulmonary complications (PPC) is considerable . The isolated effect of mobilization immediately after surgery has previously not been studied. The aim of the study is to evaluate the effects of immediate mobilization (within 2 hours after arrival to the postoperative recovery unit) after abdominal surgery and also the patients and the staffs experiences of early mobilization.

Methods: A randomized controlled trial will be conducted. A total of 300 Swedish-speaking, adult patients (≥18 years) planned for elective open or robot assisted laparascopic abdominal surgery with an expected anesthetic duration exceeding 2 hours are eligible for consecutive enrollment in the study. Patients who cannot mobilize independently before surgery, will be excluded. Procedure: Randomization to:

1. Mobilization within 2 hours after arrival to the postoperative recovery unit after surgery - to sit up as long as they can in a chair, or on the bedside + breathing exercises standardized every hour, with a PEP-device or to
2. Mobilization within 2 hours after arrival to the postoperative recovery unit after surgery - to sit up as long as they can in a chair, or on the bedside.

   or to
3. No mobilization - laying or sitting in bed with a maximum of 30° elevation of the head rest. No mobilization out of the bed or breathing exercises until discharge or a maximum of 6 hours.

Outcome assessment: The primary outcomes are arterial oxygen pressure (PaO2), and peripheral oxygen saturation (SpO2) over time and between groups. Secondary outcomes are arterial carbon dioxide pressure (PaCO2), pH, bGlu, lactate (arterial blood gas sample) over time and between groups; lung function assessed as forced vital capacity (FVC), forced expiratory flow in the one second (FEV1) and peak expiratory flow (PEF) by a micro spirometer ( preoperatively and the day after surgery); postoperative pneumonia and total length of stay at the postoperative recovery unit and at the hospital.

After the intervention both patients (n 25) and staff (n 20) will be interviewed about experiences of early mobilization.

Clinical significance: If a fairly simple and cheap intervention, such as mobilization immediately after open abdominal surgery, can lead to imporved oxygen saturation, shortened stay at hospital in total, it should be included as a routine in postoperative care.

DETAILED DESCRIPTION:
There are approximately 600 000 surgeries performed each year in Sweden. Advances in surgical technique have led to a more complex surgery on patients with more serious comorbidities. This, in turn, has led to longer operations, which expose patients to longer periods of anesthesia. During anesthesia, muscle relaxant is used, the diaphragm is then relaxed and abdominal contents are pressing against the muscle and lung tissue behind. This in combination with surgery, supine position and immobilization during a longer period of time, has a negative impact on the functional respiratory capacity (FRC) even after the surgery. The ability to cough is eliminated and produced secretion remains in the airways increasing the risk of airway closure. Therefore, the risk of postoperative pulmonary complications (PPC) such as pneumonia, atelectasis (collapsed airways in the lungs) and respiratory insufficiency, is considerable. Mobilization (to sit, stand or walk) is recomended as an intervention to improve and normalize breathing after surgery. However, the isolated effect of mobilization immediately after surgery has previously not been studied.

Hypothesis We hypothesize that immediate mobilization (within 2 hours after arrival at the postoperative recovery unit) after open or robot assisted laporascopic abdominal surgery will affect respiratory function.

Points of inquiry

1. Can mobilization or mobilization and breathing exercises (standardized every hour) with a PEP-device, at a pressure of 10-15cmH2O positive expiratory pressure (PEP) affect respiratory function ?
2. Can mobilization or mobilization and breathing exercises (PEP) reduce the prevalence of postoperative pneumonia, shorten time at the recovery unit or total length of stay at the hospital?
3. How do patients and staff expereience early mobilization after abdominal surgery?

Methods A randomized controlled trial will be conducted to evaluate whether mobilization immediately after open or robot assisted laparascopic abdominal surgery can affect respiratory function.

Patients A total of 300 Swedish-speaking, adult patients (≥18 years) planned for elective open or robot assisted laparascopic abdominal surgery with anesthetic time exceeding 2 hours at Karolinska University Hospital Solna are eligible for consecutive enrollment in the study. Patients who cannot mobilize independently before surgery will be excluded.

Procedure All patients will arrive at the postoperative recovery unit after the surgery where the randomization will take place. Patients who are considered to be in need of non-invasive ventilation immediate after the surgery, or when mobilization is contradicted due to the surgical procedure, or if they arrive to the recovery unit after 6 pm, will not be considered for randomization.

Patients will be randomized to either:

1. Mobilization within 2 hours after arrival to the postoperative recovery unit after surgery - to sit up as long as they can in a chair or on the bedside (if not possible to mobilize to a chair) + breathing exercises with a PEP-device (standardized every hour at a pressure of 10-15cmH2O) or to
2. Mobilization within 2 hours after arrival to the postoperative recovery unit after surgery - to sit up as long as they can in a chair or on the bedside (if not possible to mobilize to a chair).

   or to
3. No mobilization - that is laying in bed with a maximum of 30° elevation of the head rest. No mobilization out of the bed or breathing exercises until discharge or a maximum of 6 hours.

The study interventions will continue during 4 hours and after that all patients will receive the same treatment until they are transferred back to the surgical ward.

Data collection Baseline data such as age, sex, weight, smoking history, comorbidities, American Society of Anesthesiologists (ASA)-classification, peripheral oxygen saturation (SpO2) and results from a spirometry measurement will be collected during the meeting with the anesthesiologist at the outpatient clinic two weeks prior to surgery. Treatment- and patient care data such as need for analgesics, blood pressure, heart rate, and respiratory rate will continually be registered in a bedside case report form. Time for, duration of and frequency of mobilization will also be registered in the study protocol. Finally, information of any deaths, respiratory complications such as pneumonia, patients' length of stay at the recovery unit and at the hospital will be obtained from medical charts.

Outcome assessment The primary outcome is arterial oxygen pressure (PaO2) (kPa) (6,7), measured via arterial blood gas sample, and peripheral oxygen saturation (SpO2) , measured peripherally with a pulse oximeter PaO2 and SpO2 assessed from arrival to the postoperative recovery unit and thereafter every hour whith oxygen supply disconected for 15 minutes. Secondary outcomes are changes in arterial carbon dioxide pressure (PaCO2), ), pH, bGlu, lactate (arterial blood gas sample) over time and between groups over time and between groups; lung function assessed as forced vital capacity (FVC), forced expiratory flow in the one second (FEV1) and peak expiratory flow (PEF) by a micro spirometer (preoperatively and the day after surgery); number of patients with respiratory insufficiency, defined as SpO2 <90%, or PaO2 <8kPa and/or PaCO2 ≥6.5kPa measured without oxygen supply; postoperative pneumonia and total length of stay at the wards and at the hospital.

After the intervention both patients (n 25) and the staff (n 20) will be interviewed about their experiences of early mobilization.

Statistical analyses The number of patients required to establish a statistical power of 80% and a significance level of 5%, were 63 patients for each group. Parametric or non parametric analyses will be used depending on data level.

Clinical significance If a fairly simple and cheap intervention, such as mobilization immediately after open abdominal surgery, can lead to less postoperative complications, shortened stay at the postoperative recovery unit, and at the hospital in total, it should be included as a routine in postoperative care.

Ethical considerations The project has been approved by the Regional Ethical Review Board in Stockholm (Dnr: 2015/703-31/1, 2016/1831-32, 2016/2176-32, 2017/836-32). The patients will receive verbal and written information about the study and informed consent forms will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Swedish-speaking, adult patients (≥18 years) planned for elective open or robot assisted laparascopic abdominal surgery with anesthetic time exceeding 2 hours, at Karolinska University Hospital Solna

Exclusion Criteria:

* Patients who cannot mobilize independently before surgery will be excluded, or if not able to understand instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Arterial oxygen saturation | 1 year
  measured with blood gases
Peripheral oxygen saturation | 1 year
  measured with pulse oximetry

SECONDARY OUTCOMES:
Arterial carbon dioxide | 1 year
  measured with blood gases
pH, lactate and Bglu | 1 year
  measured with blood gases
forced vital capacity (FVC) | 1 year
  measured with spirometry
forced expiratory volume in one second (FEV1) | 1 year
  measured with spirometry
Peak expiratory flow (PEF) | 1 year
  measured with spirometry
postoperative pulmonary complications | 1 year
  Data from Medical record
Total length of stay at hospital | 1 year
  Data from Medical record

CONTACTS AND LOCATIONS:
Overall Officials: Malin Nygren-Bonnier, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svensson-Raskh A, Schandl AR, Stahle A, Nygren-Bonnier M, Fagevik Olsen M. Mobilization Started Within 2 Hours After Abdominal Surgery Improves Peripheral and Arterial Oxygenation: A Single-Center Randomized Controlled Trial. Phys Ther. 2021 May 4;101(5):pzab094. doi: 10.1093/ptj/pzab094. PMID 33742678